CLINICAL TRIAL: NCT04862247
Title: A Pilot Randomized Control Trial of a Relapse Prevention Online Exposure Protocol for Eating Disorders and Mechanisms of Change
Brief Title: Online Relapse Prevention Study
Acronym: ORP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); King's College London (Other)
Responsible Party: Principal Investigator, Cheri Levinson, Director, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#20.0626; 1R34MH124799-01 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Anorexia Nervosa, Atypical; Other Specified Feeding or Eating Disorder
Keywords: Relapse Prevention; Treatment; Eating Disorder Symptoms; Therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imaginal Exposure Condition (Experimental): Participants will complete one phone session including education about the treatment followed by four online sessions of imaginal exposure across a one month time period. Each session is separated by 1 week.
  Interventions: Behavioral: Imaginal Exposure Condition
- Writing and Thinking Condition (Active Comparator): Participants will complete one phone session including education about the treatment followed by four online sessions of a writing and thinking intervention across a one month time period. Each session is separated by 1 week.
  Interventions: Behavioral: Writing and Thinking Condition

INTERVENTIONS:
Behavioral: Imaginal Exposure Condition — Participants will be asked to think and write about an eating related fear or anxiety. Specifically, they will be asked to spend 20-30 minutes writing about a specific fear or anxiety they have, then another 20-35 minutes re-reading and imagining that what they have written is happening.
  Arms: Imaginal Exposure Condition
Behavioral: Writing and Thinking Condition — Participants will be asked to think and write about their eating disorder using specific prompts designed to help them process their eating disorder. Specifically, they will be asked to spend 20-30 minutes writing their eating disorder, then another 20-35 minutes re-reading what they wrote.
  Arms: Writing and Thinking Condition

SUMMARY:
The purpose of this study is to collect preliminary data on the feasibility and acceptability of the randomization of two relapse-prevention treatment conditions after discharge from intensive eating disorder (ED) treatment: an imaginal exposure therapy and a writing and thinking intervention. The second aim to test for (a) differences between the two treatments for the prevention of relapse and (b) preliminary change on clinical ED outcomes (e.g., ED symptoms, fears). The investigators further aim to examine the two treatments target fear extinction and if fear extinction is associated with ED outcomes. The investigators also plan to test if baseline differences in fear conditioning relate to change in ED outcomes across treatment.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* discharged from intensive treatment within the last four months (inpatient, residential, partial hospital/day program, intensive outpatient program)
* currently meet criteria for anorexia nervosa, other specified feeding and eating disorder-atypical anorexia nervosa, or bulimia nervosa

Exclusion Criteria:

* high and active suicidality, psychosis, mania, or medical compromised status will be excluded, as these comorbidities would make it difficult to complete study procedures
* under the age of 18
* does not meet criteria for anorexia nervosa, other specified feeding and eating disorder-atypical anorexia nervosa, or bulimia nervosa.
* discharged from intensive treatment more than four months ago

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Rate of Eating Disorder Relapse | 6-Month Follow-Up
  First, the investigators will define relapse as moving from one stage of remission to another (e.g., remission to partial remission or partial remission to currently ill). Second, the investigators will define relapse as re-entry into a more intensive treatment setting (e.g., moving from outpatient to partial hospitalization).
Change in Eating Disorder Symptoms using the EDE-Q | Up to 6-Month Follow-Up
  The Eating Disorder Examination Questionnaire (EDEQ), a self-reported measure, is assessed at multiple time points throughout the duration of the study and is used to examine the attitudes and behaviors in individuals with eating disorder symptoms.
Re-admission Percentage | 1 Month Follow Up and 6 Month Follow Up
  Using the Treatment Interview, we will assess all current and past treatment experiences, dates of treatment, and primary type of treatment. Re-admission will be assessed at follow up timepoints and defined as re-entry into a more intensive treatment setting.

SECONDARY OUTCOMES:
Change in State Anxiety | Treatment Session 1 through 5
  Subjective Units of Distress(SUDS) is a valid and reliable behavioral measure of state anxiety used during each treatment session to measure anxiety and distress and will be collected before, during, and after each session. Additionally, the Brief State Anxiety Measure is a 6-item measure with acceptable reliability and validity and sensitivity to fluctuations in state anxiety levels and will be collected at the beginning and end of each session.
Change in State Fear of Food | Treatment Session 2 through 5
  State Fear of Food Measure will be used to assess food anxiety, food avoidance, and feared concerns and will be collected at the beginning and end of each session.
Change in Positive and Negative Affect | Treatment Session 2 through 5
  State Positive and Negative Affect Schedule will be used to assess positive and negative affect at the beginning and end of each session.
Change in Eating Disorder Symptoms | Treatment Session 2 through 5
  Eating Disorder-15 is a 15-item measure of eating disorder cognitions and behaviors, which will be collected at the beginning of each treatment session.
Fear Extinction | Up to 6 Month Follow Up
  FLARe is a validated smart-phone behavioral assessment of fear learning that will assess target engagement at baseline, post, and one and six month follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Cheri A Levinson, PhD, Principal Investigator — University of Louisville
Locations (1):
- Eating Anxiety Treatment Laboratory and Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farrell NR, Brosof LC, Vanzhula IA, Christian C, Bowie OR, Levinson CA. [Exploring Mechanisms of Action in Exposure-Based Cognitive Behavioral Therapy for Eating Disorders: The Role of Eating-Related Fears and Body-Related Safety Behaviors]. Behav Ther. 2019 Nov;50(6):1125-1135. doi: 10.1016/j.beth.2019.01.008. Epub 2019 Feb 12. French. PMID 31735247
- [Background] Levinson CA, Brosof LC, Ma J, Fewell L, Lenze EJ. Fear of food prospectively predicts drive for thinness in an eating disorder sample recently discharged from intensive treatment. Eat Behav. 2017 Dec;27:45-51. doi: 10.1016/j.eatbeh.2017.11.004. Epub 2017 Nov 9. PMID 29145095
- [Background] Levinson CA, Christian C, Vanzhula IA. Manipulating the theoretical framing of exposure therapy for eating disorders impacts clinicians' treatment preferences. Eat Weight Disord. 2020 Oct;25(5):1205-1212. doi: 10.1007/s40519-019-00751-3. Epub 2019 Jul 17. PMID 31317512
- [Background] Murray SB, Strober M, Craske MG, Griffiths S, Levinson CA, Strigo IA. Fear as a translational mechanism in the psychopathology of anorexia nervosa. Neurosci Biobehav Rev. 2018 Dec;95:383-395. doi: 10.1016/j.neubiorev.2018.10.013. Epub 2018 Oct 28. PMID 30392878
- [Background] Reilly EE, Anderson LM, Gorrell S, Schaumberg K, Anderson DA. Expanding exposure-based interventions for eating disorders. Int J Eat Disord. 2017 Oct;50(10):1137-1141. doi: 10.1002/eat.22761. Epub 2017 Aug 16. PMID 28815659
- [Background] Levinson CA, Christian C, Ram SS, Vanzhula I, Brosof LC, Michelson LP, Williams BM. Eating disorder symptoms and core eating disorder fears decrease during online imaginal exposure therapy for eating disorders. J Affect Disord. 2020 Nov 1;276:585-591. doi: 10.1016/j.jad.2020.07.075. Epub 2020 Jul 21. PMID 32794449
- [Background] Levinson CA, Rapp J, Riley EN. Addressing the fear of fat: extending imaginal exposure therapy for anxiety disorders to anorexia nervosa. Eat Weight Disord. 2014 Dec;19(4):521-4. doi: 10.1007/s40519-014-0115-6. Epub 2014 Apr 2. No abstract available. PMID 24691784
- [Background] Steinglass JE, Sysko R, Glasofer D, Albano AM, Simpson HB, Walsh BT. Rationale for the application of exposure and response prevention to the treatment of anorexia nervosa. Int J Eat Disord. 2011 Mar;44(2):134-41. doi: 10.1002/eat.20784. PMID 20127936